CLINICAL TRIAL: NCT03678493
Title: A Randomized Placebo-Controlled Clinical Trial of Fecal Microbiota Transplantation in Patients With Acute Myeloid Leukemia and Allogeneic Hematopoietic Cell Transplantation Recipients
Brief Title: A Study of FMT in Patients With AML Allo HSCT in Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS170; MT2018-01 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia; Allogeneic Hematopoietic Cell Transplantation
Keywords: AML; Allo-HCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- AML Patients undergoing Intensive Chemotherapy (Experimental)
  Interventions: Biological: Fecal Microbiota Transplant (FMT)
- AML Patients undergoing Intensive Chemotherapy Control (Placebo Comparator)
  Interventions: Other: Placebo
- Patients undergoing Allo-HCT Patients (Experimental)
  Interventions: Biological: Fecal Microbiota Transplant (FMT)
- Patients undergoing Allo-HCT Patients Control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) — Oral Capsule
  Other Names: FMT
  Arms: AML Patients undergoing Intensive Chemotherapy; Patients undergoing Allo-HCT Patients
Other: Placebo — Oral Capsule
  Arms: AML Patients undergoing Intensive Chemotherapy Control; Patients undergoing Allo-HCT Patients Control

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial of Fecal Microbiota Transplant (FMT) in 2 independent cohorts (60 acute myeloid leukemia patients undergoing intensive chemotherapy and 60 Allo-HCT patients). Participants in each cohort will be randomized in a 2:1 ratio to receive up to 3 treatments of FMT vs. placebo after each exposure to antibacterial antibiotics until 3 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Cohort A: Patients undergoing intensive induction chemotherapy for acute myeloid leukemia (AML; newly diagnosed or relapsed/refractory).

  * Any intensive regimen with planned ~4 weeks of inpatient stay
* Cohort B: Allo-HCT patients

  * Any allogeneic transplant regimen with planned GVHD prophylaxis containing generic IV Mycophenolate Mofetil (MMF) and tacrolimus (Tac)
* Sexually active females of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control until at least six months post-FMT/placebo
* Voluntary written consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Planned continuation of antibacterial antibiotics after the first neutrophil recovery (ANC > 1,000)
* Patients who are currently receiving or recently received (within 28 days) other investigational agents.
* Pregnant or breast feeding. The FDA has not classified this agent into a specified pregnancy category. Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — University of Minnesota, Division of Hematology, Oncology and Transplantation
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Rashidi A, Ebadi M, Rehman TU, Elhusseini H, Kazadi D, Halaweish H, Khan MH, Hoeschen A, Cao Q, Luo X, Kabage AJ, Lopez S, Holtan SG, Weisdorf DJ, Khoruts A, Staley C. Randomized Double-Blind Phase II Trial of Fecal Microbiota Transplantation Versus Placebo in Allogeneic Hematopoietic Cell Transplantation and AML. J Clin Oncol. 2023 Dec 1;41(34):5306-5319. doi: 10.1200/JCO.22.02366. Epub 2023 May 26. PMID 37235836

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing Allo-HCT: Fecal Microbiota Transplant (FMT): Oral Capsule
- Patients Undergoing Allo-HCT Control: Placebo: Oral Capsule
Period: Overall Study
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
Started | 18 | 8 | 49 | 25
Completed | 18 | 8 | 49 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AML Patients Undergoing Intensive Chemothera; Patients Undergoing Allo-HCT Patients: Fecal Microbiota Transplant (FMT): Oral Capsule
- Total: Total of all reporting groups
Arm/Group | AML Patients Undergoing Intensive Chemothera | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT Patients | Patients Undergoing Allo-HCT Patients Control | Total
Number analyzed (Participants) | 18 | 8 | 49 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 7 | 31 | 22 | 74
  >=65 years | 4 | 1 | 18 | 3 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 23 | 9 | 46
  Male | 8 | 4 | 26 | 16 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 16 | 7 | 45 | 23 | 91
  Unknown or Not Reported | 2 | 1 | 2 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 3
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 15 | 8 | 45 | 23 | 91
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 8 | 49 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of FMT in AML Patients and Allo-HCT Recipients - Number of Infections
Description: Number of infections infections until 4 months after the first intervention. Monitored each visit through safety assessment.
Time Frame: 4 Months
Measure: Median (95% Confidence Interval); unit: Infections
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
Number analyzed (Participants) | 18 | 8 | 49 | 25
Infections | 1.12 [0.57 to 1.67] | 1.50 [0.35 to 2.65] | 0.89 [0.60 to 1.19] | 1.09 [0.55 to 1.64]

2. Secondary Outcome: FMT Engraftment
Description: Proportion of Donor Microbiome Fecal Microbiota Transplantation (FMT) Present in Transplant Recipient. Patient and donor samples analyzed with SourceTracker software.
Time Frame: 2 Weeks after first FMT treatment
Population: Only a subset of patients were evaluable for engraftment analysis. This is because they either didn't provide a sample or their sample didn't meet the quality criteria.
Measure: Mean (Inter-Quartile Range); unit: Proportion of Donor Microbiome FMT
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | Patients Undergoing Allo-HCT
Number analyzed (Participants) | 9 | 34
Proportion of Donor Microbiome FMT | 0.3192 [0 to .301] | 0.1117 [0 to 0.2675]

3. Secondary Outcome: FMT Engraftment
Description: as for outcome 2
Time Frame: 4 Weeks after first FMT treatment
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: Proportion of Donor Microbiome FMT
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | Patients Undergoing Allo-HCT
Number analyzed (Participants) | 1 | 18
Proportion of Donor Microbiome FMT | 0.4767 | 0.2626 [0 to 0.2452]

4. Secondary Outcome: Percentage of Participants With Grade II-IV Acute Graft-versus-host Disease (aGVHD II-IV)
Description: Percentage of Participants with Grade II-IV Acute Graft-versus-host Disease (aGVHD II-IV). Monitored each visit through safety assessment. Grade II better, Grade IV worse.
Time Frame: Day 180 post-HCT, up to 7 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Experimental: Patients Undergoing Allo-HCT: Fecal Microbiota Transplant (FMT): Oral Capsule
- Placebo Comparator: Patients Undergoing Allo-HCT Control: Placebo: Oral capsule
Arm/Group | Experimental: Patients Undergoing Allo-HCT | Placebo Comparator: Patients Undergoing Allo-HCT Control
Number analyzed (Participants) | 49 | 25
Percentage of participants | 29.8 [16.5 to 43] | 8 [0 to 19.6]

5. Secondary Outcome: Number of BSI of Suspected Gut Origin
Description: Number of BSI of suspected gut origin. Monitored each visit through safety assessment.
Time Frame: 1 week after first FMT treatment
Measure: Number; unit: Bloodstream infections
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
Number analyzed (Participants) | 18 | 8 | 49 | 25
Bloodstream infections | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Bacterial Infections
Description: Number of Bacterial Infections. Monitored each visit through safety assessment.
Time Frame: 4 Months after first FMT treatment
Measure: Number; unit: Infections
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
Number analyzed (Participants) | 18 | 8 | 49 | 25
Infections | 8 | 2 | 10 | 2

7. Secondary Outcome: Number of Viral Infections
Description: Number of Viral Infections. Monitored each visit through safety assessment.
Time Frame: 4 Months after first FMT treatment
Measure: Number; unit: Infections
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
Number analyzed (Participants) | 18 | 8 | 49 | 25
Infections | 2 | 2 | 13 | 8

8. Secondary Outcome: Number of Fungal Infections
Description: Number of Fungal Infections. Monitored each visit through safety assessment.
Time Frame: 4 Months after first FMT treatment
Measure: Number; unit: Infections
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
Number analyzed (Participants) | 18 | 8 | 49 | 25
Infections | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | AML Patients Undergoing Intensive Chemotherapy | AML Patients Undergoing Intensive Chemotherapy Control | Patients Undergoing Allo-HCT | Patients Undergoing Allo-HCT Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/8 | 6/49 | 3/25
Serious Adverse Events (participants affected / at risk) | 16/18 | 4/8 | 22/49 | 4/25
Other Adverse Events (participants affected / at risk) | 16/18 | 4/8 | 22/49 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AML Patients Undergoing Intensive Chemotherapy (N=18) | AML Patients Undergoing Intensive Chemotherapy Control (N=8) | Patients Undergoing Allo-HCT (N=49) | Patients Undergoing Allo-HCT Control (N=25)
Bloodstream infection (Infections and infestations) | 10 (10) | 2 (2) | 8 (8) | 3 (3)
Acute GVHD (Immune system disorders) | 2 (2) | 0 (0) | 9 (9) | 0 (0)
Pneumonia (Immune system disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Fever (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AML Patients Undergoing Intensive Chemotherapy (N=18) | AML Patients Undergoing Intensive Chemotherapy Control (N=8) | Patients Undergoing Allo-HCT (N=49) | Patients Undergoing Allo-HCT Control (N=25)
Bloodstream infection (Infections and infestations) | 10 (10) | 2 (2) | 8 (8) | 3 (3)
Acute GVHD (Immune system disorders) | 2 (2) | 0 (0) | 9 (9) | 0 (0)
Pneumonia (Immune system disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Fever (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03678493/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03678493/ICF_001.pdf